CLINICAL TRIAL: NCT02750735
Title: Nickel Allergy and Systemic Nickel Allergy Syndrome in Non Celiac Wheat Sensitivity
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Other Study IDs: ACPM10
Record Dates: First submitted 2016-04-15; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Non Celiac Wheat Sensitivity

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Retrospective NCWS patients: The clinical charts of NCWS patients attending the outpatient centers of the Department of Internal Medicine at the University Hospital of Palermo and the Department of Internal Medicine of the Hospital of Sciacca were retrospectively reviewed. Patients had all been diagnosed with NCWS between January 2001 and June 2011, by a DBPCC method, and included in a previously published study. These charts included specific sections for the presence of associated atopic diseases, including nickel allergy. In this way, the characteristics of the NCWS patients suffering from nickel allergy were compared with those of the NCWS patients who did not suffer from nickel allergy. Incomplete clinical charts were excluded.
- Prospective NCWS patients: The investigators also prospectively surveyed adult patients with functional gastroenterological symptoms according to the Rome III criteria, and a definitive diagnosis of NCWS. The patients were recruited between December 2014 and March 2016 at 3 centers: the two already mentioned and the Gastroenterology Unit of the ARNAS Civico Hospital of Palermo, Italy. Most of the patients had been referred due to gastrointestinal symptoms, the onset of which, they reported, could be related to wheat ingestion. Again, the characteristics of the NCWS patients suffering from nickel allergy were compared with those of the NCWS patients who did not suffer from nickel allergy.
- Retrospective NCWS control patients: To compare the frequency of nickel allergy in NCWS and non-NCWS patients, a control group composed of 70 irritable bowel syndrome (IBS) patients, was selected. These controls were randomly chosen by a computer-generated method from subjects diagnosed during the same period and age- (+/-2 years) and sex-matched (+/-5%) with the NCWS patients. The IBS controls had been receiving the same elimination diet as the NCWS patients and had not shown any clinical improvement; they belonged to the cohort of subjects the investigators had studied previously.
- Prospective NCWS control patients: As for the retrospective study, to compare the frequency of nickel allergy in NCWS and non-NCWS patients, a control group composed of 70 patients with functional gastroenterological symptoms, was selected, with the same criteria adopted for the retrospective study.

SUMMARY:
In the last few years, a new clinical entity has emerged which includes patients who consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have celiac disease (CD) or wheat allergy. This clinical condition has been named non-celiac gluten sensitivity (NCGS), although in a recent article, the investigators suggested the term "non-celiac wheat sensitivity" (NCWS), because it is not known to date what component of wheat actually causes the symptoms. Nickel is the fourth most used metal and the most frequent cause of contact allergy in the industrialized world. As a natural element of the earth's crust small amounts are found in water, soil, and natural foods, especially plant ones. Nickel allergy not only affects the skin but also results in systemic manifestations. Systemic nickel allergy syndrome can have cutaneous (urticaria/angioedema, flares, itching), and/or gastrointestinal (meteorism, colic, diarrhoea) signs and symptoms. In this study, the investigators evaluated 1) the frequency of Nickel allergy and Systemic Nickel allergy syndrome in NCWS patients, and 2) the clinical, serological, and histological characteristics of NCWS patients with contact dermatitis Nickel positive in comparison to NCWS patients without contact dermatitis.

DETAILED DESCRIPTION:
In the last few years, a new clinical entity has emerged which includes patients who consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have celiac disease (CD) or wheat allergy. This clinical condition has been named non-celiac gluten sensitivity (NCGS), although in a recent article, the investigators suggested the term "non-celiac wheat sensitivity" (NCWS), because it is not known to date what component of wheat actually causes the symptoms. Other areas of doubt in NCWS regard its pathogenesis, while some papers reported intestinal immunologic activation, others linked NCWS to the dietary short chain carbohydrate (fermentable oligo-di-monosaccharides and polyols, FODMAPs) load. The investigators recently demonstrated that higher proportions of patients with NCWS develop autoimmune disorders, are antinuclear antibodies (ANA) positive, and show DQ2/DQ8 haplotypes compared with patients with irritable bowel syndrome (IBS), supporting an immunologic involvement in NCWS. Furthermore, some papers reported also a high frequency, ranging from 22% and 35%, of coexistent atopic diseases in NCWS patients, and the investigators suggested that a percentage of NCWS patients could really suffer from non-IgE-mediated wheat allergy.

Nickel is the fourth most used metal and the most frequent cause of contact allergy in the industrialized world. As a natural element of the earth's crust small amounts are found in water, soil, and natural foods, especially plant ones. Nickel allergy not only affects the skin but also results in systemic manifestations. Systemic nickel allergy syndrome can have cutaneous (urticaria/angioedema, flares, itching), and/or gastrointestinal (meteorism, colic, diarrhoea) signs and symptoms.

Volta et al. reported that 15% of NCWS patients suffered from allergy to nickel, but they did not further characterize this subgroup of patients, neither posed the NCWS diagnosis by means the double-blind placebo controlled challenge (DBPCC), as recommended. In this study, the investigators evaluated 1) the frequency of Nickel allergy and Systemic Nickel allergy syndrome in NCWS patients, and 2) the clinical, serological, and histological characteristics of NCWS patients with contact dermatitis Nickel positive in comparison to NCWS patients without contact dermatitis.

ELIGIBILITY:
Inclusion Criteria:

All the patients met the recently proposed criteria:

* negative serum anti-tissue transglutaminase and antiendomysium (EmA) IgA and IgG antibodies;
* absence of intestinal villous atrophy;
* IgE-mediated immunoallergy tests negative to wheat (skin prick tests and/or serum specific IgE detection).

Adjunctive criteria adopted in our patients were:

* resolution of the gastrointestinal symptoms on a standard elimination diet, without wheat, cow's milk, egg, tomato, chocolate, or other food(s) causing self-reported symptoms;
* symptom reappearance on double-blind placebo-controlled (DBPC) wheat challenge, performed as described previously. As in previous studies, DBPC cow's milk protein challenge and other "open" food challenges were also performed.

Exclusion Criteria:

Exclusion criteria were:

* age < 18 years;
* positive EmA in the culture medium of the duodenal biopsies, even if the villi to crypts ratio in the duodenal mucosa was normal;
* self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study;
* other organic cutaneous and/or gastrointestinal diseases;
* concomitant treatment with steroids and/or antihistamines.

Allergic contact dermatitis was diagnosed in patients showing local eczematous lesions on the skin in close contact with nickel-containing objects. Suspected systemic nickel allergy syndrome (SNAS), was defined as a reaction characterized not only by diffused eczematous lesions (systemic contact dermatitis) but also by extracutaneous signs and symptoms, mainly gastrointestinal, after ingestion of nickel-rich foods (i.e. tomato, cocoa, beans, mushrooms, vegetables, wheat flour, etc). In all cases, the diagnosis was confirmed by means of the epicutaneous patch tests which provoked delayed lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was divided into 2 different parts. In the first, the clinical charts of NCWS patients were retrospectively reviewed, comparing the characteristics of the ones suffering from nickel allergy with those who did not suffer from nickel allergy, using, as control group, 70 IBS patients. In the second, the investigators prospectively surveyed adult patients with functional gastroenterological symptoms (Rome III criteria) and a definitive diagnosis of NCWS, comparing the characteristics of the ones suffering from nickel allergy were compared with those who did not suffer from nickel allergy, using, as control group, 70 patients with functional gastroenterological symptoms.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2001-01; Primary Completion 2011-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Nickel allergy and Systemic Nickel allergy syndrome in retrospective NCWS patients | Up to 10 years
  Frequency of Nickel allergy and Systemic Nickel allergy syndrome in retrospective NCWS patients and controls
Nickel allergy and Systemic Nickel allergy syndrome in prospective NCWS patients | Up to 15 months
  Frequency of Nickel allergy and Systemic Nickel allergy syndrome in prospective NCWS patients and controls

SECONDARY OUTCOMES:
Characteristics of retrospective NCWS patients with contact dermatitis Nickel positive in comparison to retrospective NCWS patients without contact dermatitis and controls. | Up to 10 years
  Clinical, serological, and histological characteristics of of retrospective NCWS patients with contact dermatitis Nickel positive in comparison to retrospective NCWS patients without contact dermatitis and controls.
Characteristics of prospective NCWS patients with contact dermatitis Nickel positive in comparison to prospective NCWS patients without contact dermatitis and controls. | Up to 15 months
  Clinical, serological, and histological characteristics of prospective NCWS patients with contact dermatitis Nickel positive in comparison to prospective NCWS patients without contact dermatitis and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Study Chair — University of Palermo
Locations (2):
- Italy (2):
  - Antonio Carroccio, Sciacca, Agrigento
  - Pasquale Mansueto, Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Role of FODMAPs in Patients With Irritable Bowel Syndrome. Nutr Clin Pract. 2015 Oct;30(5):665-82. doi: 10.1177/0884533615569886. Epub 2015 Feb 18. PMID 25694210
- [Background] Carroccio A, D'Alcamo A, Mansueto P. Nonceliac wheat sensitivity in the context of multiple food hypersensitivity: new data from confocal endomicroscopy. Gastroenterology. 2015 Mar;148(3):666-7. doi: 10.1053/j.gastro.2014.11.047. Epub 2015 Jan 24. No abstract available. PMID 25625764
- [Background] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Background] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Background] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Background] Carroccio A, Brusca I, Mansueto P, D'alcamo A, Barrale M, Soresi M, Seidita A, La Chiusa SM, Iacono G, Sprini D. A comparison between two different in vitro basophil activation tests for gluten- and cow's milk protein sensitivity in irritable bowel syndrome (IBS)-like patients. Clin Chem Lab Med. 2013 Jun;51(6):1257-63. doi: 10.1515/cclm-2012-0609. PMID 23183757
- [Background] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Derived] D'Alcamo A, Mansueto P, Soresi M, Iacobucci R, Blasca F, Geraci G, Cavataio F, Fayer F, Arini A, Di Stefano L, Iacono G, Bosco L, Carroccio A. Contact Dermatitis Due to Nickel Allergy in Patients Suffering from Non-Celiac Wheat Sensitivity. Nutrients. 2017 Feb 2;9(2):103. doi: 10.3390/nu9020103. PMID 28157173